CLINICAL TRIAL: NCT05801965
Title: Sidekick Health Digital Therapeutic Solution for Cancer Patients: A Feasibility Randomized Controlled Trial
Brief Title: A Digital Therapeutic Solution for Cancer Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sidekick Health (Industry)
Collaborators: Landspitali University Hospital (Other); Ljósið Cancer Rehabilitation Center (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SKH-ONC-99-003
Record Dates: First submitted 2023-03-24; First posted 2023-04-06 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2024-03

CONDITIONS: Cancer; Prostate Cancer; Colorectal Cancer; Lung Cancer
Keywords: cancer; digital solution; lifestyle change; prostate cancer; quality of life; digital intervention; side effects; medication adherence; physical activity; colorectal cancer; lung cancer
MeSH Terms: conditions — Neoplasms; Prostatic Neoplasms; Colorectal Neoplasms; Lung Neoplasms; Medication Adherence; Motor Activity | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: Single-center prospective randomized open label pilot study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Digital intervention group (Experimental): Participants will be instructed to download Sidekick Health app and receive a code to access the 14-week digital intervention in addition to standard of care, as is defined for the control arm.
  Beyond this, all participants in the interventional arm will also receive standard of care as defined for the control arm.
  Interventions: Device: A digital solution for patients with Cancer; Other: Standard of care for patients with Cancer
- Standard of care - control group (Active Comparator): Participants in the control arm will receive standard of care treatment. Standard of care includes medical treatment at Landspitali University Hospital, and optional cancer rehabilitation at the Ljósið Cancer Rehabilitation Center.
  Interventions: Other: Standard of care for patients with Cancer

INTERVENTIONS:
Device: A digital solution for patients with Cancer — A digital program that provides holistic lifestyle intervention as well as disease education.
  Other Names: SK-411 - General Oncology Program; PC-SK-451 Prostate Cancer program; CRC-SK-441; Colorectal Cancer Program LC-SK-431; Lung Cancer Program
  Arms: Digital intervention group
Other: Standard of care for patients with Cancer — Standard of care includes medical treatment at Landspitali University Hospital, and optional cancer rehabilitation at the Ljósið Cancer Rehabilitation Center.

SUMMARY:
This is a randomized, controlled trial to assess the feasibility of Sidekick Health's digital programs for cancer patients. Participants will be treated with standard of care (SoC) in combination with the digital programs, or SoC only.

We will compare the effect of the digital programs in addition to SoC to SoC only, on the cancer-related quality of life (QoL), cancer-related fatigue, and side-effect management.

DETAILED DESCRIPTION:
In line with the growing need to support cancer patients with lifestyle modifications, education and disease management, Sidekick Health developed 14-week digital programs addressing the specific needs of patients with cancers. In this study, the effect of adding the Sidekick's digital program to the standard of care (SoC) treatment for cancer patients will be assessed, with focus on prostate cancer, colorectal cancer and lung cancer. The digital programs investigated are a general oncology program (SK-411), or specific programs tailored for patients diagnosed with prostate cancer (PC-SK-451), colorectal cancer (CRC-SK-441), or lung cancer (LC-SK-431).

The study will be a single center feasibility study with an intervention group and a comparison group recruiting 84 cancer patients in active cancer treatment from Landspítali University Hospital. Patients will be randomized to receive either the SoC treatment alone or SoC with the addition of the digital program. Active cancer treatment is defined as chemotherapy, hormonal therapy, targeted therapy, immunotherapy, or radiation therapy according to standard treatment guidelines.

ELIGIBILITY:
Inclusion Criteria:

* Adults (at least 18 years of age) diagnosed with cancer
* Has started active cancer treatment (chemotherapy, hormonal therapy, targeted therapy, immunotherapy, radiotherapy) during the study
* Cancer diagnosis (all stages), with a focus on prostate cancer, lung cancer, or colorectal cancer
* Understands verbal and written Icelandic or English
* Owning a smartphone compatible with the Sidekick Health app and capable of using it.
* Capacity to give informed consent
* Willing to comply with all scheduled visits, study interventions, and procedures

Exclusion Criteria:

* Pregnancy
* Surgeries in the last 4 weeks prior to participation in the study
* Surgeries planned during the 14-weeks intervention
* Not able to comply with study intervention or scheduled measures and visits, as assessed by oncologist
* Current breast cancer diagnosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2023-04-06 (Actual); Primary Completion 2024-09-01 (Actual); Study Completion 2024-09-01 (Actual)

PRIMARY OUTCOMES:
Cancer-specific Quality of Life | Baseline, 14 , 26, and 38 weeks after inclusion in the study
  Difference in change in total score of the 30-item European Organization for the Research and Treatment of Cancer Quality of Life Questionnaire (EORTC-QLQ-C30) between the intervention and control groups.
  The EORTC-QLQ-C30 is a 30-item questionnaire. It is composed of 28 questions with a Likert scale of 4 options where 1 represents "not at all" to 4 "very much", and 2 questions with a Likert scale of 7 options where 1 represents "very poor" to 7 "excellent". Scores on the QLQ-C30 range from 30 to 126, with a lower score representing a higher quality of life.

SECONDARY OUTCOMES:
Cancer-related fatigue derived from the general cancer questionnaire subscale | Baseline, 14 , 26, and 38 weeks after inclusion in the study
  Difference in change in fatigue related subscale (questions 10, 12 and 18) of the European Organization for the Research and Treatment of Cancer Quality of Life Questionnaire (EORTC-QLQ-C30) between the intervention and control groups.
  The fatigue subscale consists of questions 10, 12, and 18 of EORTC-QLQ-C30. These 3 questions are scored on a Likert scale of 4 options where 1 represents "not at all" to 4 "very much". Scores on the fatigue subscale range from 3 to 12, with a low score representing a low level of fatigue.
Cancer-related fatigue | Baseline, 14 , 26, and 38 weeks after inclusion in the study
  Difference in change in the total score on the European Organization for the Research and Treatment of Cancer Quality of Life Questionnaire Fatigue Module (EORTC-QLQ-FA12) between the intervention and control groups.
  This 12-item questionnaire assesses physical-, cognitive- and emotional fatigue, the questionnaire is composed of 12 questions with a Likert scale of 4 options where 1 represents "not at all" to 4 "very much". Scores on the EORTC-QLQ-FA12 range from 12 to 48, with a lower score representing less fatigue.
Health-related quality of life of prostate cancer patients | Baseline, 14 , 26, and 38 weeks after inclusion in the study
  Difference in change in the scores on the European Organization for the Research and Treatment of Cancer Quality of Life Questionnaire for Prostate Cancer (EORTC-QLQ-PR25) between the prostate cancer patients in the intervention and control groups.
  The EORTC QLQ-PR25 questionnaire assesses symptoms related to prostate cancer, its treatment, and aspects of life related to this type of cancer. It consists of 25 questions with a Likert scale of 4 options where 1 represents "not at all," to 4 "very." The questions included in the questionnaire are grouped into symptom scales (questions 1 to 19) and functional scales (questions 20-25).
  For the EORTC QLQ-PR25 questionnaire, a higher score on the symptomatic scales means a greater severity of symptoms, while a higher score on question 20-22 and a lower score on questions 23-25 of the functional scales means a higher level of functioning.
Health-related quality of life of lung cancer patients | Baseline, 14 , 26, and 38 weeks after inclusion in the study
  Difference in change in the total score on the European Organization for the Research and Treatment of Cancer Quality of Life Questionnaire for Lung Cancer (EORTC-QLQ-LC13) between the lung cancer patients in the intervention and control groups.
  The EORTC-QLQ-LC13 is a 13-item questionnaire. It is composed of 13 questions with a Likert scale of 4 options where 1 represents "not at all" to 4 "very much". Scores on the EORTC-QLQ-LC13 range from 13 to 52, with a lower score representing a higher quality of life.
Health-related quality of life of colorectal cancer patients | Baseline, 14 , 26, and 38 weeks after inclusion in the study
  Difference in change in the total score on the European Organization for the Research and Treatment of Cancer Quality of Life Questionnaire for Colorectal Cancer (EORTC-QLQ-CR29) between the colorectal cancer patients in the intervention and control groups.
  The EORTC-QLQ-CR29 is a 29-item questionnaire. It is composed of 29 questions with a Likert scale of 4 options where 1 represents "not at all" to 4 "very much", with some of these questions specific for people with or without a stoma bag, and two specific questions for each sex. Scores on the EORTC-QLQ-CR29 range from 25 to 104 with a lower score (on all but one of the two specific questions for each sex) representing a higher quality of life.
Depression, anxiety, and stress levels | Baseline and 14 weeks after inclusion in the study
  Difference in change in the total score of the 21-item Depression, Anxiety and Stress Scale (DASS21) questionnaire between the intervention and control group.
  Each question has a Likert scale of 4 options where 0 represents "did not apply to me" to 3 "applied to me very much". The scores on the subscales range from 0 to 63, and low scores indicate a better mental health status.
Cancer- and treatment-specific side effects | Baseline and 14 weeks after inclusion in the study
  Evaluate the difference in cancer- and treatment-specific side effects in the intervention group between baseline and end of intervention.
  Side effects are measured through in-app patient reported outcomes (PROs): patients evaluate their symptoms, grading them on a scale of 1 to 10, where low scores indicate the mildest symptoms and high scores indicate the most severe symptoms.
Sleep, energy, and stress levels | Baseline and 14 weeks after inclusion in the study
  Evaluate the difference in sleep, energy, and stress levels in the intervention group between base line and end of intervention.
  Sleep, energy, and stress levels are measured through in-app patient reported outcomes (PROs). Patients score their sleep, energy, and stress levels, grading them on a scale of 1 to 10. Low scores indicate poor sleep quality, low energy levels, and low stress levels. High scores indicate good sleep quality, high energy levels, and stress levels.
Self-assessed health-related quality of life for health economic evaluation | Baseline, 14 , 26, and 38 weeks after inclusion in the study
  Difference in change in total score of the self-assessed EuroQuol Five Dimension - Five Level (EQ-5D-5L) health questionnaire between the intervention and control groups EQ-E5-5L scores range from -0.530 to 1, with higher scores indicating a better health status. A score of 1 indicates full health.
Patients' disease related self-efficacy | Baseline and 14 weeks after inclusion in the study
  Difference in change in a 6-item Self-Efficacy for Managing Chronic Disease questionnaire (SEMCD) score between the intervention and control groups.
  The SEMCD covers several domains that are common across many chronic diseases, such as symptom control, role function, emotional functioning, and communicating with physicians.
  The SEMCD questionnaire is composed of 6 questions with Likert scales of 10 options where 1 represents "not at all confident" to 10 "totally confident". Scores on the SEMCD range from 6 to 60, with a higher score representing a higher self-efficacy.
User satisfaction in intervention group | 14 weeks
  Scores in the mHealth App Usability Questionnaire (MAUQ) of the intervention group.
  The MAUQ is an 18-item questionnaire. It is composed of questions with Likert scales of 7 options where 1 represents "strongly disagree" to 7 "strongly agree". Scores on the MAUQ range from 18 to 126, with a higher score representing a higher usability.
User retention | 14 weeks
  Percentage of participants that will complete the digital intervention (DTx) program. Where "complete" is defined as finishing 75% of program.
User engagement | 14 weeks
  Percentage of participants that are active in the digital intervention (DTx) program. Where "active" is defined as visiting the app at least once per week.

CONTACTS AND LOCATIONS:
Locations (2):
- Iceland (2):
  - Landspitali University Hospital, Reykjavik
  - Ljósið Cancer Rehabilitation Center, Reykjavik

IPD SHARING:
Plan to Share IPD: No
Anonymized Individual Participant Data may be shared with other researchers for relevant research purposes following complementary ethical review and approval from the Ethical Review Board.